CLINICAL TRIAL: NCT00008021
Title: A Phase I Study of 90Y-DOTA-Peptide-Lym-1 With Peripheral Blood Stem Cell Support, Paclitaxel And Cyclosporin A In Patients With Non-Hodgkin's Lymphoma
Brief Title: Monoclonal Antibody Therapy, Chemotherapy, and Peripheral Stem Cell Transplantation in Treating Patients With Refractory Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Davis (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: UCD-991860; CDR0000068363 (Registry Identifier: PDQ (Physician Data Query)); NCI-V00-1638
Record Dates: First submitted 2001-01-06; First posted 2003-06-02 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2002-12

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Filgrastim; Lym-1 monoclonal antibody; Cyclosporine; Paclitaxel; Peripheral Blood Stem Cell Transplantation; Indium

INTERVENTIONS:
Biological: filgrastim
Biological: monoclonal antibody Lym-1
Drug: cyclosporine
Drug: paclitaxel
Procedure: peripheral blood stem cell transplantation
Radiation: indium In 111 monoclonal antibody Lym-1
Radiation: yttrium Y 90 monoclonal antibody Lym-1

SUMMARY:
RATIONALE: Monoclonal antibodies can locate cancer cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplantation may allow doctors to give higher doses of chemotherapy and kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibody therapy, cyclosporine, and paclitaxel followed by peripheral stem cell transplantation in treating patients who have refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of yttrium Y 90 monoclonal antibody Lym-1 administered with cyclosporine and paclitaxel followed by autologous peripheral blood stem cell transplantation in patients with refractory non-Hodgkin's lymphoma.
* Determine the toxicity of this treatment regimen in these patients.

OUTLINE: This is an open-label, dose escalation study of yttrium Y 90 monoclonal antibody Lym-1 (Y90 MOAB Lym-1). Patients are assigned to one of four cohorts.

* Cohort I: Patients receive filgrastim (G-CSF) subcutaneously (SC) beginning 4 days prior to peripheral blood stem cell (PBSC) mobilization and continuing until adequate PBSC are collected. Patients receive unlabeled monoclonal antibody (MOAB) Lym-1 IV followed by a tracer dose of indium In 111 MOAB Lym-1 (In111 MOAB Lym-1) IV on day 0 and unlabeled MOAB Lym-1 IV followed by Y90 MOAB Lym-1 IV on day 7. Patients also receive oral cyclosporine every 12 hours on days -2 to 14. Patients may undergo autologous PBSC transplantation, if necessary, no earlier than day 17 and receive G-CSF SC beginning at the completion of PBSC re-infusion and continuing until blood counts recover.
* Cohort II: Patients undergo PBSC mobilization and receive treatment as in cohort I. Patients also receive paclitaxel IV over 3 hours on day 9.
* Cohort III: Patients undergo PBSC mobilization and receive unlabeled MOAB Lym-1, In111 MOAB Lym-1, Y90 MOAB Lym-1, and cyclosporine as in cohort I and paclitaxel as in cohort II. Patients undergo autologous PBSC transplantation no earlier than day 17. Patients receive G-CSF after transplantation as in cohort I.
* Cohort IV: Patients undergo PBSC mobilization and receive treatment as in cohort III. Treatment repeats every 6 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 1 to 3 patients receive escalating doses of Y90 MOAB Lym-1 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 1 of 3 patients require PBSC transplantation, or the dose preceding that at which 2 of 3 patients experience dose-limiting toxicity.

Patients are followed monthly for 3 months, every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A maximum of 40 patients will be accrued for this study within 36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-Hodgkin's lymphoma (NHL) that has failed standard therapy

  * Any grade allowed
  * Intermediate or high grade NHL must have failed standard therapy with curative intent
* Measurable disease
* HAMA titer negative
* NHL tissue Lym-1 reactive in vitro
* Bilateral bone marrow biopsy less than 25% NHL
* No evidence of myelodysplastic syndrome in bone marrow NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 130,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST no greater than 84 U/L

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* LVEF at least 50%

Pulmonary:

* FEV1 at least 60% of predicted
* FVC at least 60% of predicted
* Corrected DLCO at least 50%

Other:

* No other malignancy within the past 5 years except for non- melanoma skin cancer
* HIV negative
* No AIDS
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy involving more than 25% of bone marrow
* At least 4 weeks since prior external beam radiotherapy

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-02

CONTACTS AND LOCATIONS:
Overall Officials: Gerald L. DeNardo, MD, Study Chair — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States